CLINICAL TRIAL: NCT02680899
Title: Adolescent Outcomes in Mental Health InSciEd Out
Brief Title: Adolescent Mental Health InSciEd Out
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Christopher Pierret, Assistant Professor of Biochemistry and Molecular Biology, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 15-009107
Record Dates: First submitted 2016-02-02; First posted 2016-02-12 (Estimated); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Mental Disorders; Substance-Related Disorders; Social Stigma; Mental Health Wellness 1; Mental Health Impairment
Keywords: science education; health promotion; mental health promotion; stigmatization; behavioral intervention
MeSH Terms: conditions — Mental Disorders; Substance-Related Disorders; Social Stigma; Stereotyping

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Curricular Intervention (Experimental): The intervention is a novel science education curriculum in mental health and addiction called My Mind, My Body.
  Interventions: Behavioral: Curricular Intervention

INTERVENTIONS:
Behavioral: Curricular Intervention — The intervention is a novel grades 7 and 8 InSciEd Out curriculum in mental health and addiction called My Mind, My Body.

SUMMARY:
The study herein seeks to determine whether students undergoing InSciEd Out curriculum in mental health and addiction (called My Mind, My Body) experience changes in their mental health-related knowledge, attitudes, and help-seeking behavioral intentions. The research group hypothesizes that students undergoing InSciEd Out mental health and addiction curriculum will exhibit pre-post increases in mental health literacy, decreases in mental health stigmatization, and increases in mental health help-seeking behavioral intentions.

DETAILED DESCRIPTION:
Integrated Science Education Outreach (InSciEd Out) is one novel program that seeks to promote scientific and health literacy through fostering scientific inquiry. The guiding premise of InSciEd Out's health promotion arm is a concept called Prescription Education (PE), which uses science education as a direct and early intervention for disease behaviors. The underlying hypothesis of InSciEd Out PE is that a student who lives a scientific experience in his or her own voice (undergoes true inquiry-based science) will be empowered to elect healthier behaviors in any targeted health paradigm. PE's proposed mechanism of change is that inquiry-based science catalyzes transitions from knowledge to understanding to attitudes to intents to actual behavioral change.

InSciEd Out partnership with the the school in this study began in Spring of 2013 with a projected health promotion arm targeting mental health and addiction. The current iteration of the partnership commenced in Summer of 2014 under the annual InSciEd Out summer internship. This internship led to creation of grades 7 and 8 curriculum in mental health and addiction. Version 1 of this curriculum was piloted last year. A revised version of the curriculum will be implemented in Spring of 2016. Although there are education-specific metrics for assessment already built into program evaluation of InSciEd Out, there are currently no clinically relevant inventories in place to specifically probe efficacy of the lesson plans upon key mental health outcomes.

The study herein is the establishment of clinically relevant inventories around implemented InSciEd Out curriculum in mental health and addiction (called My Mind, My Body). These inventories are selected to measure student changes in their mental health-related knowledge, attitudes, and help-seeking behavioral intentions. The research group hypothesizes that students undergoing InSciEd Out mental health and addiction curriculum will exhibit pre-post increases in mental health literacy, decreases in mental health stigmatization, and increases in mental health help-seeking behavioral intentions.

ELIGIBILITY:
Inclusion Criteria: Partner school students who do not opt out of and assent to the study

Exclusion Criteria: Partner school students opting out of or not assenting to the study

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-02; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Score on General Help-Seeking Questionnaire at 1 month | Baseline and then at study completion, estimated to be ~1 month
  The general help-seeking questionnaire: vignette version (GHSQ-V) will be used to assess help-seeking behavioral intentions.
Change from Baseline Score on Westbrook Mental Health Knowledge Test at 1 month | Baseline and then at study completion, estimated to be ~1 month
  The Westbrook Knowledge Test assesses mental health knowledge.
Change from Baseline Score on Adolescent Attribution Questionnaire at 1 month | Baseline and then at study completion, estimated to be ~1 month
  The adolescent attribution questionnaire (AQ-8-C) will be used to assess mental illness stigmatization.

SECONDARY OUTCOMES:
Teacher Report of Student Outcomes | Conducted at study completion, estimated to be ~1 month
  Teacher quotes from semi-structured interviews concerning student outcomes in mental health knowledge, attitudes, and behaviors will be used to form a student narrative.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Pierret, PhD, Principal Investigator — Mayo Clinic; Stephen C Ekker, PhD, Principal Investigator — Mayo Clinic; Joanna Yang, BS, Study Director — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang J, Lopez Cervera R, Tye SJ, Ekker SC, Pierret C. Adolescent mental health education InSciEd Out: a case study of an alternative middle school population. J Transl Med. 2018 Apr 3;16(1):84. doi: 10.1186/s12967-018-1459-x. PMID 29615090